CLINICAL TRIAL: NCT03149120
Title: Phase II Randomized Study of Nivolumab With or Without Pazopanib in Metastatic or Unresectable Soft Tissue Sarcomas After One Prior Line of Systemic Therapy or Ineligible to Receive an Anthracycline-based Treatment
Brief Title: Study of Nivolumab With or Without Pazopanib in Metastatic or Unresectable Soft Tissue Sarcomas
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: No patient enrolled as new similar study will be in system within 3 months
Sponsor: NYU Langone Health (Other)
Collaborators: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 16-02078
Record Dates: First submitted 2017-04-27; First posted 2017-05-11 (Actual); Last update posted 2017-08-22 (Actual); Status verified 2017-08

CONDITIONS: Soft Tissue Sarcomas
Keywords: Metastatic; Unresectable; anthracycline; chemotherapy; systemic therapy
MeSH Terms: conditions — Sarcoma; Neoplasm Metastasis | interventions — Nivolumab; pazopanib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Nivolumab (Experimental): Nivolumab will be given as an intravenous infusion at a dose of 240 mg every 2 weeks for at least 6 months.
  Interventions: Biological: Nivolumab
- Nivolumab with Pazopanib (Experimental): Pazopanib at a dose of 800mg by mouth daily.
  Interventions: Biological: Nivolumab; Drug: Pazopanib

INTERVENTIONS:
Biological: Nivolumab — Nivolumab will be given as an intravenous infusion at a dose of 240 mg every 2 weeks for at least 6 months.
  Other Names: Opdivo
Drug: Pazopanib — Pazopanib given at a dose of 800 mg by mouth daily.
  Other Names: Votrient
  Arms: Nivolumab with Pazopanib

SUMMARY:
This trial will assess whether nivolumab alone or nivolumab combined with pazopanib will be associated with an improvement in progression free survival (PFS) at 6 months

DETAILED DESCRIPTION:
The investigators hypothesize that the nivolumab alone or nivolumab plus pazopanib will be associated with an improvement in progression free survival (PFS) at 6 months compared to historical controls of placebo and pazopanib alone respectively.

This is a randomized, Phase 2 study of nivolumab alone or nivolumab plus pazopanib in adult (≥ 18 years old) male and female subjects with unresectable or metastatic soft tissue sarcoma either ineligible to receive an anthracycline-based first line treatment or after one prior systemic therapy. Up to 33 and 46 subjects will be randomized (1:1) in the nivolumab and nivolumab plus pazopanib cohorts respectively, with a Simon two-stage design. Preliminary endpoint analysis will be performed when at least 18 subjects in the nivolumab cohort and 16 subjects in the nivolumab plus pazopanib cohort, have completed the first 12 cycles of nivolumab (6 months). Accrual duration is expected to be around 2 years.

ELIGIBILITY:
Inclusion Criteria:

* Histologic diagnosis of metastatic or unresectable soft tissue or bone sarcoma
* No prior therapy with nivolumab in either cohorts or with pazopanib in the combination cohort
* At least one line of systemic therapy or ineligibility for an anthracycline based chemotherapy
* At least 2 distinct measurable metastatic sites
* Adequate organ and marrow function as defined by initial laboratory tests
* Life expectancy > 3 months
* Stable brain metastases for at least 4 weeks and no steroid dependence

Exclusion Criteria:

* Autoimmune disease Any underlying medical or psychiatric condition, which in the opinion of the Investigator, will make the administration of study drugs hazardous or obscure the interpretation of adverse events
* Concomitant therapy with any non-study immunotherapy regimens, cytotoxic chemotherapy, immunosuppressive agents, other investigation therapies Chronic use of systemic corticosteroids greater than prednisone 10 mg daily or its equivalent
* Women of childbearing potential who are unwilling or unable to use an acceptable method to avoid pregnancy for the entire study period and for at least 5 months after cessation of study drug, or have a positive pregnancy test at baseline, or are pregnant or breastfeeding;
* Prisoners or subjects who are compulsorily detained (involuntarily incarcerated) for treatment of either a psychiatric or physical illness.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2017-08 (Estimated); Primary Completion 2017-08-17 (Actual); Study Completion 2022-06 (Estimated)

PRIMARY OUTCOMES:
Progression-free survival (PFS) at 6 months for nivolumab alone or nivolumab in combination with pazopanib | 6 Months
  Time from randomization until disease progression or death

SECONDARY OUTCOMES:
Measure of Tolerability | 6 Months
  Time from randomization to disease progression, death, or discontinuation of treatment for any reason (eg, toxicity, patient preference, or initiation of a new treatment without documented progression)
Overall Response Rate | 6 Months
  Proportion of patients with reduction in tumor burden of a predefined amount
Median Progression Free Overall Survival (OS) | 6 Months
  Time from randomization until death from any cause

CONTACTS AND LOCATIONS:
Overall Officials: Luca Paoluzzi, Principal Investigator — NYU Langone Health
Locations (1):
- New York University School of Medicine, New York, New York, United States